CLINICAL TRIAL: NCT02635893
Title: Lower Limb Function After Spinal Cord Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Monica Perez, Chair Arms + Hands Lab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20150605
Record Dates: First submitted 2015-12-11; First posted 2015-12-21 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Spinal Cord Injury
Keywords: SCI
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- D-Cycloserine/Placebo + Stimulation (Active Comparator): Participant will be given a single dose of 100 mg of D-Cycloserine or placebo before receiving stimulation.
  Interventions: Drug: D-Cycloserine; Drug: Placebo; Other: Stimulation
- Training+Med/Placebo+Stimulation (Active Comparator): Participant will be given a single dose of 100 mg of D-Cycloserine or placebo before receiving stimulation followed by training.
  Interventions: Drug: D-Cycloserine; Drug: Placebo; Other: Training; Other: Stimulation
- Training+Med+Stimulation/Placebo Stim (Active Comparator): Participant will be given a single dose of 100 mg of D-Cycloserine or placebo before receiving stimulation or placebo stimulation followed by training.
  Interventions: Drug: D-Cycloserine; Other: Training; Other: Stimulation; Other: Placebo Stimulation

INTERVENTIONS:
Drug: D-Cycloserine — 100 mg of Seromycin by mouth will be administered
  Other Names: Seromycin
Drug: Placebo — placebo pill will be administered instead of medication by mouth
  Other Names: Placebo Drug
  Arms: D-Cycloserine/Placebo + Stimulation; Training+Med/Placebo+Stimulation
Other: Training — walking around a designated track at different speeds both forward and backward
  Arms: Training+Med+Stimulation/Placebo Stim; Training+Med/Placebo+Stimulation
Other: Stimulation — magnetic stimulation and electrical stimulation may be applied
Other: Placebo Stimulation — this is a fake stimulation that is administered but will be unknow to the subject.
  Arms: Training+Med+Stimulation/Placebo Stim

SUMMARY:
This is a randomized, experimental study that examines the physiology of central nervous system pathways contributing to the control of bilateral movements in individuals with spinal cord injuries and promotes the recovery of lower-limb motor function through the use of stimulation and locomotor training.

DETAILED DESCRIPTION:
This study plans to examine plasticity in corticospinal synapses of lower-limb muscles. it has been demonstrated that plasticity elicited at corticospinal synapses in the spinal cord result in enhancements in electromyographic (EMG) and force activity in upper-limb muscles. The first step in this proposal is to determine if synaptic plasticity can be elicited in corticospinal projections targeting lower-limb muscles in humans with SCI.

We will also study methods to strengthen corticospinal plasticity to promote recovery of leg clearance during training. We will use two novel strategies to enhance plasticity in corticospinal synapses of lower-limb muscles after SCI: a). administration of an N-methyl-D-aspartate (NMDA) receptor agonist (i.e. D-cycloserine), and b). Combine NMDA-induced corticospinal plasticity with training (2D lower limb training and locomotor training. Corticospinal synaptic plasticity is thought to depend on activation of NMDA receptors and D-cycloserine enhances motor skill behaviors in animals and humans will be enhanced by NMDA-induced corticospinal plasticity. An important strength of this aim is the combination of training and strategies that aimed at enhancing the synaptic efficacy of residual corticospinal projections. Training effects on physiological pathways will be explored and correlated with locomotor function

ELIGIBILITY:
Inclusion Criteria:

* 4. Inclusion criteria for individuals with SCI:

  * Male and females between ages 18-85 years of age
  * SCI ( ≥1 month of injury)
  * ASIA A, B,C and D
  * SCI above L5
  * Able to perform a visible contraction with dorsiflexor and hip flexor muscles (allowing testing of largely impaired patients)
  * Able to ambulate a few steps with or without an assistive device

Inclusion criteria for healthy controls:

* Male and females between ages 18-85 years of age
* Able to walk and complete lower-limb tests with both legs

Exclusion Criteria:

Exclusion criteria for individuals with SCI

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease,
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke,
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants.
* Pregnant females, and
* Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida or herniated cervical disk.

Exclusion criteria for healthy controls:

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease,
* Any debilitating disease that causes exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke,
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants.
* Pregnant females, and
* Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida or herniated cervical disk.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-04-11 (Actual)

PRIMARY OUTCOMES:
Changes in motor evoked potential size | 30 minutes before and 30 minutes after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Perez, PT, Phd, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- The Shirley Ryan Ability Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No